CLINICAL TRIAL: NCT00608712
Title: Use Of Esomeprazole In Postoperative Bariatric Surgery Patients Users And Non-Users Of Nonsteroidal Anti-Inflammatory Drugs (NSAIDS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D9612L00097
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Postoperative Bariatric Surgery
Keywords: bariatric surgery; ulcer prevention
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 20mg oral tablet
  Other Names: Nexium

SUMMARY:
Phase IV, open-label, multicenter, non-randomized, with 2 non-comparative investigational arms study, carried out in morbid obesity patients who had undergone gastric bypass surgery for body weight reduction

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated
* BMI ≥40 kg/m2 or BMI between 35 and 40 kg/m2, but with a severe disease together with obesity
* Indication for gastric bypass surgery
* Upper digestive endoscopy prior to surgery not showing esophagitis, erosions, ulcers or neoplasia, examination performed up to 30 days before surgery being considered valid
* Helicobacter pylori non-infected patients, diagnosed by tests carried out up to 30 days before surgery

Exclusion Criteria:

* Contraindication for gastric bypass surgery
* Contraindication to use Omeprazole and derivatives
* Patients carriers of gastrinoma or having hypergastrinemia
* Patients contraindicated to perform UDE
* Patients with previous esophagogastroduodenal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Esomeprazole in preventing anastomotic stomal ulcer after gastric bypass surgery for weight loss

SECONDARY OUTCOMES:
To evaluate the efficacy of Esomeprazole in avoiding appearance of related peptic acid symptoms after gastric bypass surgery for weight loss.